CLINICAL TRIAL: NCT00889070
Title: Respiratory Events Among Premature Infants (32-<36 w/GA) - Outcomes & Risk Tracking Study (The REPORT Study)
Brief Title: Respiratory Events Among Premature Infants
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Hanaa Elhefni, MD, MS, MPH, MedImmune LLC
Other Study IDs: MI-MA192
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Respiratory Syncytial Virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Stage 1 (Pilot Study) All infants enrolled in the pilot stage and completing baseline screening will be evaluated as the analyzable set.

SUMMARY:
Assess the burden of disease associated with RSV infection with premature children in an outpatient setting.

DETAILED DESCRIPTION:
The primary objective of this prospective study is to assess the burden of disease associated with RSV infection, as measured/determined by rates of outpatient medically attended LRI, emergency room visits and hospitalization among preterm infants (32-≤36 wGA) during RSV season, and its medical/health consequences, as measured by wheezing events, the infant's first RSV season, up to May 2009.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent/guardian to participate in study
* Male or female preterm infants 32-≤36 wGA
* Infant is ≤ 6month old at the time of enrollment
* Parent/guardian has the ability and willingness to follow study protocol (during the first RSV season) as required by the protocol

Exclusion Criteria:

* Receipt of any RSV prophylactic agent: palivizumab, IGIV, or motavizumab at any time prior to enrollment
* Participation in trials of investigational RSV prophylaxis or RSV therapeutic agents
* Presence of BPD or CHD (other than surgically treated PDA, ASD or VSD)
* Condition that limits life span to 6 months or less from the date of enrollment

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male or female preterm infants 32-≤36 wGA
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The rate of RSV positivity and rate of outpatient and/or inpatient LRI events as well as the rate of outpatient and inpatient wheezing events. | Seasonal: 2008-09

SECONDARY OUTCOMES:
Evaluate characteristics of infants in RSV risk factor and rate and reason of attrition. | Seasonal: 2008-09

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa Elhefni, MD, MS, MPH, Study Director — MedImmune LLC
Locations (5):
- United States (5):
  - Children's Primary Care Medical Group, Inc., San Diego, California
  - North Florida Pediatrics, Lake City, Florida
  - Woburn Pediatric Associates, Woburn, Massachusetts
  - Suny Upstate Medical University, Syracuse, New York
  - Senders Pediatrics, Cleveland, Ohio